CLINICAL TRIAL: NCT06152575
Title: A PHASE 3, OPEN-LABEL STUDY OF ELRANATAMAB MONOTHERAPY VERSUS ELOTUZUMAB, POMALIDOMIDE, DEXAMETHASONE (EPd) OR POMALIDOMIDE, BORTEZOMIB, DEXAMETHASONE (PVd) OR CARFILZOMIB, DEXAMETHASONE (Kd) IN PARTICIPANTS WITH RELAPSED/REFRACTORY MULTIPLE MYELOMA WHO RECEIVED PRIOR ANTI-CD38 DIRECTED THERAPY
Brief Title: MagnetisMM-32: A Study to Learn About the Study Medicine Called Elranatamab in People With Multiple Myeloma (MM) That Has Come Back After Taking Other Treatments (Including Prior Treatment With an Anti-CD38 Antibody and Lenalidomide)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C1071032; MAGNETISMM-32 (Other: Alias Study Number); 2023-507871-23-00 (Registry Identifier: CTIS (EU))
Expanded Access: Available
Record Dates: First submitted 2023-11-17; First posted 2023-11-30 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Multiple Myeloma
Keywords: Elranatamab; B-Cell Maturation Antigen; BCMA; Bispecific antibody; BCMA-CD3 bispecific antibody; Myeloma; Multiple myeloma; Relapsed multiple myeloma; Refractory multiple myeloma; MagnetisMM; MagnetisMM-32; Pomalidomide; Elotuzumab; Bortezomib; Carfilzomib; PF-06863135
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — elotuzumab; pomalidomide; Dexamethasone; Bortezomib; carfilzomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Elranatamab (Experimental): Participants will receive elranatamab monotherapy
  Interventions: Drug: Elranatamab
- Investigator's Choice (Active Comparator): Participants will receive either Elotuzumab, Pomalidomide and Dexamethasone (EPd), or Pomalidomide, Bortezomib and Dexamethasone (PVd), or Carfilzomib and Dexamethasone (Kd)
  Interventions: Drug: Elotuzumab; Drug: Pomalidomide; Drug: Dexamethasone; Drug: Bortezomib; Drug: Carfilzomib

INTERVENTIONS:
Drug: Elranatamab — Elranatamab will be administered subcutaneously
  Arms: Elranatamab
Drug: Elotuzumab — Elotuzumab will be administered intravenously
  Arms: Investigator's Choice
Drug: Pomalidomide — Pomalidomide will be administered orally
  Arms: Investigator's Choice
Drug: Dexamethasone — Dexamethasone will be administered orally
  Arms: Investigator's Choice
Drug: Bortezomib — Bortezomib will be administered subcutaneously or intravenously
  Arms: Investigator's Choice
Drug: Carfilzomib — Carfilzomib will be administered intravenously
  Arms: Investigator's Choice

SUMMARY:
The purpose of this study is to learn about the study medicine called elranatamab.This study aims to compare elranatamab to other medicines for the treatment of MM (a type of cancer).

This study is seeking participants who:

* Are 18 years of age or older and have MM.
* Have received treatments before for MM.
* Have MM that has returned or not responded to their most recent treatment.

Half of the participants will receive elranatamab. The other half of participants will receive a combination therapy selected by the study doctor. The selected combination therapy will include 2 to 3 different medicines commonly used to treat MM.

Elranatamab will be given as a shot under the skin at the study clinic about once a week. This may change to a smaller number of shots later in the study.

The medicines in the combination therapy will be taken by mouth (at home or at the study clinic) AND will be given either as:

* a shot under the skin at the study clinic
* through a needle in the vein at the study clinic The number of times these medicines will be taken depends on what combination therapy the study doctor selects.

Participants may continue to receive elranatamab or a combination therapy until their MM is no longer responding. The study team will see how each participant is doing with the study treatment during regular visits at the study clinic. The study team will continue to follow-up with participants after study treatment with telephone contacts (or visits).

The study will compare the experiences of people receiving elranatamab to those people receiving a combination therapy. This will help learn about the safety and how effective elranatamab is.

ELIGIBILITY:
Inclusion Criteria:

* Prior diagnosis of multiple myeloma as defined by International Myeloma Working Group (IMWG) criteria and previously received 1 to 4 prior lines of therapy including prior anti-cluster of differentiation 38 (CD38) antibody and prior lenalidomide.
* Documented evidence of progressive disease or failure to achieve a response to last line of therapy per IMWG criteria.
* Measurable disease defined as at least 1 of the following: (a) Serum M-protein ≥0.5 g/dL; (b) Urinary M-protein excretion ≥200 mg/24 hours; (c) Serum involved immunoglobulin FLC ≥10 mg/dL AND abnormal serum immunoglobulin kappa to lambda FLC ratio (<0.26 or >1.65).
* Have clinical laboratory values within the specified range.
* ECOG (Eastern Cooperative Oncology Group) performance status ≤2.
* Not pregnant or breastfeeding and willing to use contraception.

Exclusion Criteria:

* Smoldering multiple myeloma.
* Plasma cell leukemia.
* Amyloidosis.
* Polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy and skin abnormalities (POEMS) syndrome.
* Known central nervous system (CNS) involvement or clinical signs of myelomatous meningeal involvement.
* Stem cell transplant within 12 weeks prior to enrolment, or active graft versus host disease.
* Any active, uncontrolled bacterial, fungal, or viral infection.
* Any other active malignancy within 3 years prior to enrolment (exceptions include, adequately treated basal cell or squamous cell skin cancer, carcinoma in situ)
* Previous treatment with a B cell maturation antigen (BCMA)-directed therapy or CD3-redirecting therapy.
* Unable to receive investigator's choice therapy.
* Live attenuated vaccine within 4 weeks of the first dose of study intervention.
* Administration with an investigational product (e.g. drug or vaccine) within 30 days preceding the first dose of study intervention used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 492 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival per International Myeloma Working Group criteria | Up to approximately 5 years
  From date of randomization to date of progressive disease, discontinuation from study, death, or censoring, whichever occurs first

SECONDARY OUTCOMES:
Overall survival | Up to approximately 5 years
  From date of randomization to date of discontinuation from study, death, or censoring, whichever occurs first
Progression free survival on next-line treatment per International Myeloma Working Group criteria | Up to approximately 5 years
  From date of randomization to date of second objective disease progression, discontinuation from the study, death, or censoring, whichever occurs first
Objective response rate per International Myeloma Working Group criteria | Up to approximately 5 years
  From date of randomization to date of progressive disease, discontinuation from study, death, or start of new anticancer therapy
Duration of response per International Myeloma Working Group criteria | Up to approximately 5 years
  From date of confirmed objective response to date of progressive disease, discontinuation from study, death, or censoring, whichever occurs first
Very good partial response or better response rate per International Myeloma Working Group criteria | Up to approximately 5 years
  From date of randomization to date of progressive disease, discontinuation from study, death, or start of new anticancer therapy, whichever occurs first
Complete response rate per International Myeloma Working Group criteria | Up to approximately 5 years
  From date of randomization to date of progressive disease, discontinuation from study, death, or start of new anticancer therapy, whichever occurs first
Duration of complete response per International Myeloma Working Group criteria | Up to approximately 5 years
  From date of confirmed complete response to date of progressive disease, discontinuation from study, death, or censoring, whichever occurs first
Time to response per International Myeloma Working Group criteria | Up to approximately 5 years
  From date of randomization to date of confirmed objective response
Minimal residual disease negativity rate per International Myeloma Working Group criteria | Up to approximately 5 years
  From date of randomization to date of progressive disease, discontinuation from study, death, or start of new anticancer therapy, whichever occurs first
Sustained minimal residual disease negativity rate per International Myeloma Working Group criteria | Up to approximately 5 years
  From date of randomization to date of progressive disease, discontinuation from study, death, or start of new anticancer therapy, whichever occurs first
Duration of minimal residual disease negativity rate per International Myeloma Working Group criteria | Up to approximately 5 years
  From date of minimal residual disease negativity to date of relapse, death, or censoring, whichever occurs first
Frequency of treatment-emergent adverse events | From date of first dose of study intervention up to 90 days after last study intervention administration
Frequency of abnormal laboratory results | From date of first dose of study intervention up to 90 days after last study intervention administration
Free elranatamab serum trough concentration [Ctrough] | From date of first dose of elranatamab up to approximately 14 days after last dose of elranatamab
Elranatamab immunogenicity by anti-drug antibodies against elranatamab | From date of first dose of elranatamab up to approximately 14 days after last dose of elranatamab
Health-related quality of life by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 | From date of informed consent up to approximately 35 days after last administration of study intervention
  Change from baseline scores
Health-related quality of life by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Myeloma 20 | From date of informed consent up to approximately 35 days after last administration of study intervention
  Change from baseline scores

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (265):
- United States (81):
  - Infirmary Cancer Care, Mobile, Alabama
  - Western Regional Medical Center, Inc. dba. City of Hope Phoenix, Goodyear, Arizona
  - Beverly Hills Cancer Center, Beverly Hills, California
  - Community Cancer Institute, Clovis, California
  - Clinical Research Advisors (Encino Satellite Location), Encino, California
  - Hoag Health Center Irvine, Irvine, California
  - Hoag Hospital Irvine, Irvine, California
  - Clinical Research Advisors (Korea Town Satellite Location), Los Angeles, California
  - Clinical Research Advisors (West Hollywood Satellite Location), Los Angeles, California
  - Valkyrie Clinical Trials, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Mission Community Hospital (Satellite Site), Panorama City, California
  - University of California Davis (UC Davis) Comprehensive Cancer Center, Sacramento, California
  - University of California, Sacramento, California
  - UCHealth Poudre Valley Hospital, Fort Collins, Colorado
  - UCHealth Harmony, Fort Collins, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - UCHealth Longs Peak Hospital, Longmont, Colorado
  - UCHealth Longs Peak Medical Center, Longmont, Colorado
  - UCHealth - Medical Center of the Rockies, Loveland, Colorado
  - Sylvester Comprehensive Cancer Center - The Lennar Foundation Medical Center, Coral Gables, Florida
  - University of Miami Hospital and Clinics - Deerfield Beach, Deerfield Beach, Florida
  - Sylvester Comprehensive Cancer Center- Doral, Doral, Florida
  - Sylvester Comprehensive Cancer Center - Hollywood, Hollywood, Florida
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - University of Miami Hospital and Clinics - Griffin Cancer Research Building, Miami, Florida
  - University of Miami Hospital and Clinics, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Sylvester Comprehensive Cancer Center- Kendall, Miami, Florida
  - BRCR Global, Plantation, Florida
  - BRCR Global - Tamarac, Tamarac, Florida
  - Endeavor Health - Swedish Hospital, Chicago, Illinois
  - Endeavor Health - Evanston Hospital, Evanston, Illinois
  - Endeavor Health - Glenbrook Hospital Ambulatory Care Center, Glenview, Illinois
  - Endeavor Health - Highland Park Hospital Health Center 1, Highland Park, Illinois
  - Simmons Cancer Institute at SIU, Springfield, Illinois
  - Springfield Clinic Main Campus, Springfield, Illinois
  - HSHS St. John's Hospital, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Midwestern Regional Medical Center, Inc. dba City of Hope Chicago, Zion, Illinois
  - Community Health Network, Inc., Indianapolis, Indiana
  - American Oncology Partners, P.A. Dba MidAmerica Cancer Care, Kansas City, Kansas
  - Ascentist Doctors' Hospital, Leawood, Kansas
  - American Oncology Partners, P.A. Dba MidAmerica Cancer Care, Merriam, Kansas
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - BIDMC Research Pharmacy, Boston, Massachusetts
  - American Oncology Partners, P.A. Dba MidAmerica Cancer Care, Belton, Missouri
  - MIVA Medical, Independence, Missouri
  - Kansas City VA Medical Center, Kansas City, Missouri
  - American Oncology Partners, P.A. Dba MidAmerica Cancer Care, Kansas City, Missouri
  - Bryan Medical Center, Lincoln, Nebraska
  - NHO Revive Research Institute, LLC, Lincoln, Nebraska
  - Atlantic Health System Morristown Medical Center, Morristown, New Jersey
  - WMCHealth Advanced Physician Services, Hawthorne, New York
  - Northwell Health/ RJ Zuckerberg Cancer Center, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Westchester Medical Center, Valhalla, New York
  - Brody school of Medicine at East Carolina University, Greenville, North Carolina
  - ECU Health Medical Center, Greenville, North Carolina
  - Sanford Fargo Medical Center, Fargo, North Dakota
  - Oncology Hematology Care Clinical Trials, LLC, Cincinnati, Ohio
  - TriHealth Cancer Institute-Good Samaritan Hospital, Cincinnati, Ohio
  - The Jewish Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - AHN West Penn Hospital, Pittsburgh, Pennsylvania
  - Brown University Health Cancer Institute, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island
  - St Francis Cancer Center, Greenville, South Carolina
  - Baylor University Medical Center, Investigational Drug Services, Department of Pharmacy, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Houston Methodist Willowbrook Hospital, Houston, Texas
  - US Oncology Investigational Products Center (IPC), Irving, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas
  - Baylor Scott & White Medical Center - Temple, Temple, Texas
  - West Virginia University, Morgantown, West Virginia
  - University of Wisconsin Carbone Cancer Center-University Hospital, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Clinical Science Center, Madison, Wisconsin
- Argentina (4):
  - Instituto Alexander Fleming, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Hospital Universitario Austral, Pilar, Buenos Aires
  - Hospital Italiano de Buenos Aires, Ciudad de Buenos Aires, Buenos Aires F.D.
  - Hospital Italiano de La Plata, La Plata
- Australia (7):
  - Blacktown Hospital, Blacktown, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - St Vincent's Hospital (Melbourne), Fitzroy, Victoria
  - Barwon Health, Geelong, Victoria
  - Sir Charles Gairdner Hospital, Haematology Clinical Trials, Nedlands, Western Australia
- Belgium (7):
  - Clinique Saint Pierre, Ottignies, Brabant Wallon
  - UZ Brussel, Brussels, Bruxelles-capitale, Région de
  - Grand Hôpital de Charleroi, Gilly, Hainaut
  - Centre Hospitalier Epicura, Hornu, Hainaut
  - CHR Verviers - La Tourelle, Verviers, Liège
  - Université Catholique de Louvain-Namur - Centre Hospitalier Universitaire Dinant-Godinne - Site Godi, Yvoir, Namur
  - AZ Delta vzw, Roeselare, West-vlaanderen
- Brazil (19):
  - Instituto D'Or de Pesquisa e Ensino (IDOR) - Filial Salvador, Salvador, Estado de Bahia
  - Instituto Oncomed de Educação e Pesquisa, Niterói, Rio de Janeiro
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Centro Gaucho Integrado De Oncologia, Hematologia, Ensino E Pesquisa, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisa Clínica - Área Administrativa, Porto Alegre, Rio Grande do Sul
  - Hospital Mae de Deus, Porto Alegre, Rio Grande do Sul
  - Hospital Amaral Carvalho, Jaú, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo (USP), Ribeirão Preto, São Paulo
  - Instituto D'Or de Pesquisa e Ensino (IDOR), São Paulo, São Paulo
  - Clínica Médica São Germano LTDA, SP, São Paulo
  - Instituto de Educação, Pesquisa e Gestão em Saúde, Rio de Janeiro
  - Americas Centro de Oncologia Integrado, Rio de Janeiro
  - ESHO Empresa de Serviços Hospitalares S.A/ Hospital Samaritano de Higienópolis, São Paulo
  - Instituto D'Or de Pesquisa e Ensino (IDOR), São Paulo
  - Hospital do Coracao, São Paulo
  - HU UNIFESP / SPDM - Hospital São Paulo, São Paulo
  - Universidade Federal de Sao Paulo, São Paulo
  - INSUMA, São Paulo
  - Clínica Médica São Germano S/S Ltda, São Paulo
- Canada (3):
  - The Moncton Hospital, Moncton, New Brunswick
  - Jewish General Hospital, Montreal, Quebec
  - Centre intégré universitaire de santé et de services sociaux du Nord-de-l'Île-de-Montréal (CIUSSS NÎ, Montreal, Quebec
- Chile (4):
  - FALP, Santiago, Santiago Metropolitan
  - Clínica Inmunocel, Santiago, Santiago Metropolitan
  - Clínica Universidad de Los Andes, Santiago, Santiago Metropolitan
  - Clínica Alemana de Santiago, Santiago, Santiago Metropolitan
- Croatia (7):
  - Klinicki bolnicki centar Osijek, Osijek
  - Klinicki bolnicki centar Rijeka, Rijeka
  - Klinicki bolnicki centar Split, Split
  - Sestre milosrdnice University Hospital Center, Zagreb
  - University Hospital Center Zagreb, Zagreb
  - Klinicka bolnica Dubrava, Zagreb
  - Klinicka bolnica Merkur, Zagreb
- Czechia (3):
  - Fakultní nemocnice Brno Bohunice, Brno, Brno-město
  - Fakultni nemocnice Olomouc, Olomouc, Olomoucký kraj
  - Fakultni nemocnice Kralovske Vinohrady, Prague, Praha 10
- Denmark (3):
  - Rigshospitalet, Copenhagen, Capital Region
  - Aarhus Universitetshospital, Skejby, Aarhus, Central Jutland
  - Aalborg Universitetshospital, Syd, Aalborg, North Denmark
- Finland (5):
  - Oulun yliopistollinen sairaala, Oulu, North Ostrobothnia
  - Kuopion Yliopistollinen Sairaala, Kuopio, Northern Savonia
  - Tampereen yliopistollinen sairaala, Tampere, Pirkanmaa
  - Turku University Hospital, Turku, Southwest Finland
  - Helsinki University Hospital - Comprehensive Cancer Center (HYKS - Syöpäkeskus), Helsinki, Uusimaa
- France (17):
  - CHU Bordeaux Haut-Leveque, Pessac, Aquitaine
  - Institut Universitaire du Cancer Toulouse - Oncopole - CHU de TOULOUSE, Toulouse, Haute-garonne
  - Centre Hospitalier de Dunkerque, Dunkirk, Hauts-de-France
  - Centre Hospitalier Régional Universitaire de Nancy - Hôpitaux de Brabois, Vandœuvre-lès-Nancy, Lorraine
  - Centre Hospitalier Universitaire de Nantes - L' Hopital l'hôtel-Dieu, Nantes, Pays de la Loire Region
  - Hôpital NOVO, Cergy-Pontoise, Val-d'oise
  - Hôpital NOVO, Pontoise, Val-d'oise
  - Henri Mondor Hospital, Créteil, Val-de-marne
  - CHD Vendee, La Roche-sur-Yon, Vendée
  - Centre Hospitalier Universitaire de Poitiers, Poitiers, Vienne
  - Centre Hospitalier de la Côte Basque, Bayonne
  - Centre Hospitalier du Mans, Le Mans
  - Hôpital Universitaire Necker Enfants Malades, Paris
  - Hopitaux Universitaires Paris Centre-Hopital Cochin, Paris
  - Centre Hospitalier de Cornouaille, Quimper
  - Centre Hospitalier Régional Universitaire de Tours - Hôpital Bretonneau, Tours
  - Centre Hospitalier Bretagne Atlantique, Vannes
- Germany (11):
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Robert Bosch Krankenhaus GmbH, Stuttgart, Baden-Wurttemberg
  - Universitaetsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Klinikum Nürnberg Nord, Nuremberg, Bavaria
  - Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Universitätsklinikum Jena, Jena, Thuringia
  - Vivantes Klinikum Am Urban, Berlin
  - Medizinische Universität Lausitz - Carl Thiem, Cottbus
  - Asklepios Altona, Hamburg
  - St. Barbara-Klinik Hamm-Heessen, Hamm
  - Diakonissen-Stiftungs-Krankenhaus Speyer, Speyer
- Greece (6):
  - University General Hospital of Alexandroupoli, Alexandroupoli, Anatolikí Makedonía KAI Thráki
  - Evangelismos General Hospital of Athens, Athens, Attikí
  - Alexandra General Hospital of Athens, Athens, Attikí
  - "Theagenio" Cancer Hospital of Thessaloniki, Thessaloniki, Kentrikí Makedonía
  - G. Papanikolaou General Hospital, Thessaloniki, Thessaloníki
  - University Hospital of Ioannina, Ioannina, Ípeiros
- Israel (5):
  - Rabin Medical Center, Petah Tikva, Central District
  - Sheba Medical Center, Ramat Gan, Central District
  - Hadassah Medical Center, Jerusalem, Jerusalem
  - Soroka Medical Center, Beersheba, Southern District
  - Sourasky Medical Center, Tel Aviv, TELL ABĪB
- Italy (11):
  - IRCCS - Istituto Romagnolo per lo Studio dei Tumori (IRST) "Dino Amadori", Meldola, Emilia-Romagna
  - P.O. San Carlo Borromeo- ASST SANTI PAOLO E CARLO, Milan, Lombardy
  - Azienda Socio Sanitaria Ovest milanese, Legnano, Milano
  - Azienda Ospedaliero-Universitaria Città della Salute e della Scienza di Torino, Turin, Piedmont
  - A.O.U. Policlinico Paolo Giaccone, Palermo, Sicily
  - Azienda Ospedaliero Universitaria delle Marche, Ancona, The Marches
  - Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Tuscany
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola, Bologna
  - Istituto Europeo di Oncologia IRCCS, Milan
  - Ospedale Civile dello Spirito Santo, Pescara
- Japan (17):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Toyohashi Municipal Hospital, Toyohashi, Aichi-ken
  - Ehime Prefectural Central Hospital, Matsuyama, Ehime
  - Ogaki Municipal Hospital, Ōgaki, Gifu
  - Gunma University Hospital, Maebashi, Gunma
  - National Hospital Organization Shibukawa Medical Center, Shibukawa, Gunma
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Iwate Medical University Hospital, Shiwa-gun Yahaba-cho, Iwate
  - Shizuoka Cancer Center, Nagaizumi-cho, Shizuoka
  - Nippon Medical School Hospital, Bunkyo-ku, Tokyo
  - Japanese Foundation for Cancer Research, Koto, Tokyo
  - Yamanashi Prefectural Central Hospital, Kofu, Yamanashi
  - Kagoshima University Hospital, Kagoshima
  - University Hospital,Kyoto Prefectural University of Medicine, Kyoto
  - National Hospital Organization Okayama Medical Center, Okayama
  - Okayama Rosai Hospital, Okayama
  - Yamagata University Hospital, Yamagata
- Netherlands (3):
  - Maastricht UMC+, Maastricht, Limburg
  - Albert Schweitzer Ziekenhuis, locatie Dordwijk, Dordrecht, South Holland
  - Erasmus Medisch Centrum, Rotterdam, South Holland
- Norway (4):
  - Akershus Universitetssykehus, Lørenskog, Akershus
  - St. Olavs Hospital, Trondheim, Sør-trøndelag
  - Sykehuset i Vestfold, Tønsberg, Vestfold
  - Oslo Universitetssykehus Ullevål, Oslo
- Portugal (4):
  - Instituto Português de Oncologia de Lisboa Francisco Gentil, Lisbon, Lisbon District
  - 2Ca Braga, Braga
  - Unidade Local de Saúde de Coimbra, E.P.E., Coimbra
  - Hospital da Luz Lisboa, Lisbon
- Slovakia (5):
  - Fakultna nemocnica s poliklinikou F.D.Roosevelta Banska Bystrica, Banská Bystrica, Banská Bystrica Region
  - Univerzitna Nemocnica L. Pasteura Kosice, Košice, Košice Region
  - Narodny onkologicky ustav, Bratislava
  - Univerzitna nemocnica Bratislava, Nemocnica sv. Cyrila a Metoda, Bratislava
  - Univerzitna nemocnica Martin, Martin, Žilina Region
- University Medical Centre Ljubljana, Ljubljana, Slovenia
- South Korea (3):
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [seoul]
- Spain (14):
  - Institut Català d'Oncologia (ICO) - Badalona, Badalona, Barcelona [barcelona]
  - Hospital Universitari Mutua Terrassa, Terrassa, Barcelona [barcelona]
  - OSI Ezkerraldea-Enkarterri-Cruces - Hospital Universitario Cruces, Barakaldo, Basque Country
  - Hospital Clínic de Barcelona, Barcelona, Catalunya [cataluña]
  - Hospital General Universitario Morales Meseguer, Murcia, Galicia [galicia]
  - Institut Català d'Oncologia (ICO) - Girona, Girona, Girona [gerona]
  - Hospital Universitario Infanta Leonor, Madrid, Madrid, Comunidad de
  - ASCIRES ECG Médica S.L, Valencia, Valenciana, Comunitat
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - H.R.U Málaga - Hospital General, Málaga
  - Centro de Diagnóstico y Resonancia Magnética, Salamanca
  - Hospital Universitario de Salamanca - Complejo Asistencial Universitario de Salamanca, Salamanca
  - Hospital Universitari i Politecnic La Fe, Valencia
- Sweden (2):
  - Falu Lasarett, Falun
  - Universitetssjukhuset Örebro, Örebro, Örebro LÄN [se-18]
- Taiwan (2):
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
- United Kingdom (17):
  - Milton Keynes Hospital, Milton Keynes, Buckinghamshire
  - Glan Clwyd Hospital, Bodelwyddan, Denbighshire [SIR Ddinbych Gb-ddb]
  - Royal Bournemouth Hospital, Bournemouth, Dorset
  - Poole Hospital, Poole, Dorset
  - Eastbourne District General Hospital, Eastbourne, EAST Sussex
  - Worthing Hospital, Worthing, EAST Sussex
  - Queen Elizabeth Hospital Birmingham, Birmingham, England
  - Maidstone Hospital, Maidstone, KENT
  - St Bartholomew's Hospital, London, London, CITY of
  - Guy's & St Thomas' NHS Foundation Trust, London, London, CITY of
  - King's College Hospital, London, London, CITY of
  - Hammersmith Hospital, London, London, CITY of
  - Churchill Hospital, Oxford, Oxfordshire
  - Royal Stoke University Hospital, Stoke-on-Trent, Staffordshire
  - Royal Marsden Hospital (Sutton), London, Sutton
  - Kent and Canterbury Hospital, Canterbury
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C1071032
- See also: MagnetisMM-32 — https://www.pfizerclinicaltrials.com/nct06152575-multiple-myeloma-trial